CLINICAL TRIAL: NCT02772120
Title: Comparison of Vaginal Progesterone Gel (Crinone 8%®) and Intramuscular Progesterone in Vitrified-Warmed Blastocyst Transfer Cycles
Brief Title: Comparison of Vaginal and Intramuscular Progesterone in Vitrified-warmed Blastocyst Transfer Cycles
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Before enrollment, suspended due to changing insurance coverage of study drugs.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elena Hesina Yanushpolsky, MD, Assistant Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWH2016progRCT
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: Infertility; In vitro fertilization; Embryo transfer; Blastocyst; Progesterone; Crinone
MeSH Terms: conditions — Infertility | interventions — Crinone; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal progesterone gel (Crinone® 8%) (Active Comparator): Crinone® 8% (90 mg of micronized progesterone in a bioadhesive vaginal gel contained in a single use, one piece applicator) is administered once 5 days prior to embryo transfer, then twice per day until the pregnancy test is negative or until the 10th week of pregnancy.
  Interventions: Drug: Vaginal progesterone gel (Crinone® 8%)
- Intramuscular Progesterone (Active Comparator): Progesterone-25 mg intramuscularly once 5 days prior to embryo transfer, then 50 mg once per day until the pregnancy test is negative or until the 10th week of pregnancy.
  Interventions: Drug: Intramuscular Progesterone

INTERVENTIONS:
Drug: Vaginal progesterone gel (Crinone® 8%) — Crinone® 8% (90 mg of micronized progesterone in a bioadhesive vaginal gel contained in a single use, one piece applicator) is administered once 5 days prior to embryo transfer, then twice per day until the pregnancy test is negative or until the 10th week of pregnancy.
  Other Names: vaginal progesterone; Crinone
  Arms: Vaginal progesterone gel (Crinone® 8%)
Drug: Intramuscular Progesterone — Progesterone-25 mg intramuscularly once 5 days prior to embryo transfer, then 50 mg once per day until the pregnancy test is negative or until the 10th week of pregnancy.
  Other Names: progesterone
  Arms: Intramuscular Progesterone

SUMMARY:
The aim of this study is to test the hypothesis that the pregnancy rates of women (ages 18-50 years) undergoing transfer of vitrified-warmed blastocysts (frozen at less than 41 years of age) as part of their IVF treatment are not different with respect to the administration of progesterone (Crinone® 8% vaginal gel versus intramuscular progesterone).

DETAILED DESCRIPTION:
The hypothesis of this study is that the type of progesterone administered (intramuscular progesterone or Crinone® 8% vaginal gel) does not affect implantation and clinical pregnancy rates in women receiving cryo-thawed blastocysts that were produced using their own eggs and frozen before age 41 years. Both intramuscular progesterone (25-100 mg compounded in oil) or vaginal progesterone (Crinone® 8% vaginal progesterone gel) are widely used for luteal phase support in patients receiving vitrified-warmed embryos. Crinone® 8% is FDA approved for progesterone supplementation or replacement as part of an Assisted Reproductive Technology (ART) treatment for infertile women with progesterone deficiency (FDA approval letter, 1997).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient age at time of embryo freezing: 18 to 40.9 years
* Patient age at embryo transfer: 18 to 50 years (i.e. women currently ages 18-50 years who are transferring embryos created using eggs retrieved from women aged 18-40.9 years)
* Blastocysts frozen by vitrification at Brigham and Women's Hospital
* Standard eligibility criteria for blastocyst transfer at Brigham and Women's Hospital

Exclusion Criteria:

* Fresh or cleavage-stage embryo transfer planned
* Gestational carrier cycles
* Natural and modified natural cycles
* Embryos frozen more than once or derived from thawed oocytes
* Embryos frozen at centers other than Brigham and Women's Hospital
* Embryos frozen using techniques other than vitrification (i.e. slow frozen)
* Patients with recurrent pregnancy loss, defined as failure of 3 or more clinical pregnancies
* Uterine factor infertility: Asherman's, submucosal fibroids, polyp greater than 1 cm at time of embryo transfer, uninterrupted hydrosalpinx
* Patients with three prior failed embryo transfers (fresh or frozen)
* BMI<18 or >40 kg/m2 at screening
* Currently breast feeding or pregnant
* Embryo biopsy performed
* Current smoking, alcohol or illicit drug use
* Allergy to study drugs
* Refusal or inability to adhere to study protocol
* Participation in other experimental drug trials concurrently within the past 60 days

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5-6 weeks
  Percentage of patients with intrauterine gestational sac by ultrasound

SECONDARY OUTCOMES:
Implantation rate | 5-6 weeks
  Maximum number of gestational sacs divided by total number of embryos transferred
Sustained implantation rate | 7 weeks
  maximum number of fetal heartbeats divided by total number of embryos transferred
Biochemical pregnancy | 6 weeks
  Positive serum b-hCG (above 5 IU/L) without subsequent ultrasound evidence of pregnancy
Ongoing pregnancy rate | 7-8 weeks
  Live intrauterine pregnancy at the time of transfer to obstetrical care

CONTACTS AND LOCATIONS:
Overall Officials: Elena Yanushpolsky, MD, Principal Investigator — Assistant Professor, Harvard Medical School, Director of Reproductive Surgery at Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, He Y, Zhao X, Ji X, Hong Y, Wang Y, Zhu Q, Xu B, Sun Y. Crinone Gel for Luteal Phase Support in Frozen-Thawed Embryo Transfer Cycles: A Prospective Randomized Clinical Trial in the Chinese Population. PLoS One. 2015 Jul 29;10(7):e0133027. doi: 10.1371/journal.pone.0133027. eCollection 2015. PMID 26222435
- [Background] Lightman A, Kol S, Itskovitz-Eldor J. A prospective randomized study comparing intramuscular with intravaginal natural progesterone in programmed thaw cycles. Hum Reprod. 1999 Oct;14(10):2596-9. doi: 10.1093/humrep/14.10.2596. PMID 10527993
- [Background] Shapiro DB, Pappadakis JA, Ellsworth NM, Hait HI, Nagy ZP. Progesterone replacement with vaginal gel versus i.m. injection: cycle and pregnancy outcomes in IVF patients receiving vitrified blastocysts. Hum Reprod. 2014 Aug;29(8):1706-11. doi: 10.1093/humrep/deu121. Epub 2014 May 20. PMID 24847018
- [Background] Berger BM, Phillips JA. Pregnancy outcomes in oocyte donation recipients: vaginal gel versus intramuscular injection progesterone replacement. J Assist Reprod Genet. 2012 Mar;29(3):237-42. doi: 10.1007/s10815-011-9691-9. Epub 2012 Feb 4. PMID 22310935
- See also: Drug information for progesterone — http://druginfo.nlm.nih.gov/drugportal/name/Progesterone